CLINICAL TRIAL: NCT03892590
Title: Anaylsis of Gut Microbiota in ICU
Brief Title: Gut Microbiota Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Armed Forces Goyang Hospital (Other Government)
Responsible Party: Principal Investigator, Maru Kim, Dr., The Catholic University of Korea
Other Study IDs: Gut Microbiota
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Microbiota; Metabolism
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable patient: Stable patients who admitted to ICU for observation.
  Interventions: Biological: Gut microbiota

INTERVENTIONS:
Biological: Gut microbiota — Status of microbiota

SUMMARY:
Microbiota is known to effect metabolism. This is pilot study to get status of microbiota from normal control. It will be compared to data from specific patients in ICU via further study.

DETAILED DESCRIPTION:
Microbiota is known to effect metabolism. Patients in specific conditions like hypovolemic shock, sepsis might have changes in status of microbiota. This is pilot study to get status of microbiota from normal control. Stable patient who are admitted to ICU for observation will be gathered. Samples will be collected via rectal swab at time of admission and analyzed via Next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years old
* Every patients who are admitted to ICU

Exclusion Criteria:

* With history of disease such as cancer, Crohn's disease, ulcerative colitis, irritable bowel syndrome
* With history of immunosuppressive agents.
* Initial systolic blood pressure <100
* Initial pulse rate > 100
* Need emergent operation at brain or torso
* Need vasopressor, transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable adult patient who are admitted to ICU
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Normal microbiota | 1day
  Status of microbiota of stable patient in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Maru Kim, MD, PhD, Study Chair — The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No